CLINICAL TRIAL: NCT04848844
Title: The PAtients pResenTing With COngenital HeaRt DIseAse Register (ARTORIA-R): A Global Register to Investigate Factors Associated With Morbidity and Mortality in Adult Patients With Congenital Heart Disease (ACHD) on the Waiting List for Heart or Heart/Lung Transplantation
Brief Title: The PAtients pResenTing With COngenital HeaRt DIseAse Register (ARTORIA-R)
Acronym: ARTORIA-R
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Collaborators: Deutsches Zentrum für Herz-Kreislauf-Forschung (DZHK) (Other)
Responsible Party: Sponsor
Other Study IDs: 2023-101119-BO-ff
Record Dates: First submitted 2021-04-07; First posted 2021-04-19 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Congenital Heart Disease; Heart Failure; Transplant; Complication, Failure; Arrythmia; Ventricular Dysfunction
MeSH Terms: conditions — Heart Defects, Congenital; Heart Failure; Arrhythmias, Cardiac; Ventricular Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patient transplanted due to ACHD and heart failure: Patients successfully transplanted due to congenital heart failure.
- ACHD listed due to heart failure for heart or heart and combined organ transplantation: Patients on the actual waiting list for heart or heart and combined organ transplantation. They can have either outcome transplantation or the primary outcome death on the waiting list or delisting due to clinical worsening. The secondary outcome is as well delisting due to clinical improvement.
- ACHD evaluated for heart transplantation: All patients evaluated for heart or heart and combined organ transplantation at the hospital level

SUMMARY:
Advances in surgical and medical care have led to improved outcomes in patients with congenital heart disease (CHD). As a consequence, the majority of patients nowadays survives to adulthood (adults with CHD, that is, adult CHD [ACHD]) with good quality of life. Despite the surgical success, the morbidity and mortality of ACHD is higher than in the general population and is linked to the development of heart failure (HF) in adulthood.

HF occurs in approximately 25% of patients with ACHD, even in those patients in whom the congenital mal-formation has been corrected successfully in childhood. The time course and presentation are heterogeneous owing to variable congenital malformation and limitation of treatment options. ACHD with an anatomic right ventricle as the systemic ventricle (e.g., atrial switch operation in patients with transposition of the great arteries [TGAs]) and those with a functional single ventricle (e.g., Fontan circulation) appear to be at higher risk of developing HF. Young age at initial corrective surgery-often in the ﬁrst 2 years of life-and lack of speciﬁc medical therapies can contribute to a high and early demand for heart transplantation in patients with ACHD.

DETAILED DESCRIPTION:
The ARTORIA-R is an international, observational research project collecting retrospective data from 18 countries in the period 1989 to 2024 and will thereafter include data prospectively (Figure 1). These data include patient profiles at time of evaluation for listing, listing, waiting list dynamics, post-transplant data and basic donor data. Future data will be updated annually in July each year and each institution willing to contribute anonymised data to the register is invited to participate. Furthermore, the institutions and organ allocation agencies have to obtain a positive vote of the ethic committee responsible for the data transmission of anonymized patient data.

The inclusion criteria are: a. The patient has to be listed as an adult transplant candidate in the country the data is obtained with an age ≥18 years b. The patient has to have a congenital heart defect or an inherited cardiomyopathy (specific; hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy or non-compaction cardiomyopathy) which is often included into the category ACHD c. Data is obtained from the first evaluation for listing or listing for heart-only or heart-combined organ transplantation d. Transfer of anonymised data e. The institution/organization agrees to the memorandum how data is managed, and scientific cooperation is planned between all institutions. The registry has the aim to achieve meticulous information regarding the underlying congenital heart defect and the previous treatment of the patient. With these information the patients can be divided into different cohorts with a systemic left ventricle, a systemic right ventricle or a single ventricle (which can be either an anatomic left or right ventricle). Further data is acquired regarding the medical treatment, the haemodynamic evaluation of the patient, laboratory testing to assess additional organ function of the kidney or liver, treatment in the intermediate care or intensive care unit. As it is of special relevance in ACHD patient treatment of arrhythmia, antiarrhythmic medication and use of ICD or cardiac resynchronization therapy are evaluated. Were available the data regarding imaging at listing with ejection fraction for the systemic ventricle with echocardiography or cardiac magnetic resonance imaging are obtained.

The exclusion criteria is: a. The patient is listed for a second heart transplantation (retransplantation) During the ongoing study additional institutions and organizations will be asked to include their data as well. Although the initial data is retrospective additional data into the register will be entered prospectively.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has to be listed as an adult transplant candidate in the country the data is obtained with an age ≥18 years
2. The patient has to have a congenital heart defect or an inherited cardiomyopathy (specific; hypertrophic cardiomyopathy, arrhythmogenic right ventricular cardiomyopathy or non-compaction cardiomyopathy) which is often included into the category ACHD
3. Data is obtained from the first evaluation for listing or listing for heart-only or heart-combined organ transplantation
4. Transfer of anonymised data
5. The institution/organization agrees to the memorandum how data is managed, and scientific cooperation is planned between all institutions

Exclusion Criteria:

a. The patient is listed for a second heart transplantation (retransplantation)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The PAtients pResenTing with COngenital HeaRt DIseAse Register (ARTORIA-R) will collect data from patients with ACHD evaluated or listed for heart or heart-combined organ transplantation from 19 countries in Europe and the Asia/Pacific region. We plan retrospective collection of data from 1989 - 2024 and will include patients prospectively. The primary outcome is the combined endpoint of delisting due to clinical worsening or death on the waiting list. The secondary outcome is delisting due to clinical improvement while on the waiting list.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-09-02 (Actual); Primary Completion 2030-07-30 (Estimated); Study Completion 2030-07-30 (Estimated)

PRIMARY OUTCOMES:
Delisting due to clinical worsening or death on the waiting list | Baseline: The data will be entered into the study database and afterwards during follow-up each year the status of the patient is updated
  If the patients has a clinical worsening of their status due to advanced heart failure he or she is removed from the waiting list. Patients can as well die while on the waiting list as a consquence of heart failure

SECONDARY OUTCOMES:
Delisting due to clinical improvement | Baseline: The data will be entered into the study database and afterwards during follow-up each year the status of the patient is updated
  Patients can improve from the status at listing and can be removed from the waiting list due to clinical improvement of their clinical status and not fulfilling the criteria for listing for heart or heart and combined organ transplantation anymore.

OTHER OUTCOMES:
All-cause mortality following transplantation | Baseline: The data will be entered into the study database and afterwards during follow-up each year the status of the patient is updated
  When a patient was succesfully transplanted and receives follow-up visits at the transplant center. The patient status of being alive is noted.
Implantation of a ventricular assist device as a bridge to transplantation or candidacy. Some of the patients will receive the ventricular assiste device as well as destination therapy | Baseline: The data will be entered into the study database and afterwards during follow-up each year the status of the patient is updated
  Patient is successfully treated with a ventricular assist device as a bridge to transplantation or candidacy. Some patients will receive the device as well as destination therapy

CONTACTS AND LOCATIONS:
Overall Officials: Christoph Sinning, MF, Principal Investigator — University Heart & Vascular Center Hamburg
Locations (1):
- University Heart and Vascular Center Hamburg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: Yes
Data is shared with investigators participating in the register and provide patient data to the register
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The data base is shared with the researchers institution on demand. The researcher will receive a password protected copy of the study data base. The data base only includes anonymized data.

REFERENCES:
- [Background] Sinning C, Zengin E, Diller GP, Onorati F, Castel MA, Petit T, Chen YS, Lo Rito M, Chiarello C, Guillemain R, Coniat KN, Magnussen C, Knappe D, Becher PM, Schrage B, Smits JM, Metzner A, Knosalla C, Schoenrath F, Miera O, Cho MY, Bernhardt A, Weimann J, Gossling A, Terzi A, Amodeo A, Alfieri S, Angeli E, Ragni L, Napoleone CP, Gerosa G, Pradegan N, Rodrigus I, Dumfarth J, de Pauw M, Francois K, Van Caenegem O, Ancion A, Van Cleemput J, Milicic D, Moza A, Schenker P, Thul J, Steinmetz M, Warnecke G, Ius F, Freyt S, Avsar M, Sandhaus T, Haneya A, Eifert S, Saeed D, Borger M, Welp H, Ablonczy L, Schmack B, Ruhparwar A, Naito S, Hua X, Fluschnik N, Nies M, Keil L, Senftinger J, Ismaili D, Kany S, Csengeri D, Cardillo M, Oliveti A, Faggian G, Dorent R, Jasseron C, Blanco AP, Marquez JMS, Lopez-Vilella R, Garcia-Alvarez A, Lopez MLP, Rocafort AG, Fernandez OG, Prieto-Arevalo R, Zatarain-Nicolas E, Blanchart K, Boignard A, Battistella P, Guendouz S, Houyel L, Para M, Flecher E, Gay A, Epailly E, Dambrin C, Lam K, Ka-Lai CH, Cho YH, Choi JO, Kim JJ, Coats L, Crossland DS, Mumford L, Hakmi S, Sivathasan C, Fabritz L, Schubert S, Gummert J, Hubler M, Jacksch P, Zuckermann A, Laufer G, Baumgartner H, Giamberti A, Reichenspurner H, Kirchhof P. Study design and rationale of the pAtients pResenTing with cOngenital heaRt dIseAse Register (ARTORIA-R). ESC Heart Fail. 2021 Dec;8(6):5542-5550. doi: 10.1002/ehf2.13574. Epub 2021 Sep 12. PMID 34510806
- [Background] Becher PM, Schrage B, Weimann J, Smits J, Magnussen C, Reichenspurner H, Gossling A, Rodrigus I, Dumfarth J, de Pauw M, Francois K, van Caenegem O, Ancion A, Van Cleemput J, Milicic D, Moza A, Schenker P, Rohrich L, Schonrath F, Thul J, Steinmetz M, Schmack B, Ruhparwar A, Warnecke G, Rojas SV, Sandhaus T, Haneya A, Eifert S, Welp H, Ablonczy L, Wagner F, Westermann D, Bernhardt AM, Knappe D, Blankenberg S, Kirchhof P, Zengin E, Sinning C. Clinical characteristics and outcomes of patients with adult congenital heart disease listed for heart and heart-lung transplantation in the Eurotransplant region. J Heart Lung Transplant. 2020 Nov;39(11):1238-1249. doi: 10.1016/j.healun.2020.07.012. Epub 2020 Jul 25. PMID 32778365